CLINICAL TRIAL: NCT06792656
Title: Forest Therapy for International Students
Brief Title: Measuring the Effectiveness of Forest Therapy to Alleviate Stress Among International Students
Acronym: FTIS-2024
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Nature and Forest Therapy Alliance (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: QA/109559/VICBH-2024-438742
Record Dates: First submitted 2025-01-16; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Stress Disorders; Stress; Anxiety; Anxiety Depression (Mild or Not Persistent); Sleep Deprivation; Sleep Disorders, Circadian Rhythm; Stress, Psychological; Lack of Physical Activity
Keywords: Forest Therapy; Public health; stress; nature-connectedness
MeSH Terms: conditions — Stress Disorders, Traumatic; Anxiety Disorders; Lymphoma, Follicular; Sleep Deprivation; Sleep Disorders, Circadian Rhythm; Stress, Psychological; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 2-hrs standardized Forest Therapy session (Experimental): the intervention follows the strict protocol (script) of the INFTA Forest Therapy Guiding Sequence
  Interventions: Other: standardized Forest Therapy session (120 min)

INTERVENTIONS:
Other: standardized Forest Therapy session (120 min) — standardized, 2-hrs Forest Therapy session following the INFTA Forest Therapy Guiding Sequence

SUMMARY:
International students often face high levels of stress, leading to mental health conditions, from factors including cultural and social change, educational system, financial insecurity and family responsibilities. Barriers in seeking support for mental health include stigmatisation and high costs. Single psychotherapy sessions are often unaffordable and pharmaceuticals are often associated with adverse side effects having limited efficacy.

Hence, alternative approaches and therapies are needed to manage students' wellbeing. Forest Therapy offers a low-risk lifestyle activity, which is beneficial to physical and mental health through nature exposure and increased social connection.

Thus, this research project aims to investigate to which degree guided Forest Therapy sessions may help to prevent or alleviate stress among international students in Victoria. Free Forest Therapy sessions will be offered to international students at the Royal Botanic Gardens Melbourne which is centrally located and can easily be reached by foot, car, bike or Public transport. The sessions will be offered at different dates/times during August, September and October 2024. Next to participating in the guided Forest Therapy sessions, brief surveys will be administered before and after each session which are optional.

DETAILED DESCRIPTION:
1. Eligibility

   All international students currently studying, planning to study of having completed their studies at a university in Victoria (Melbourne or regional) are eligible and invited to participate.

   Participation in this research project is voluntary.
2. Details and Proceedings

   Forest Therapy is an evidence-based Public health practice involving a complementary blend of simple physical and mental activities, undertaken in a forested surroundings. Guided Forest Therapy sessions help participants to slow down and activate their senses while enjoying walking mindfully through nature.

   All Forest Therapy sessions will take place at the Royal Botanic Gardens Melbourne (Birdwood Avenue, Melbourne 3004 VIC) and start/end at its Visitor Centre. Facilities are available at the Visitor Centre as well as throughout the Botanic Gardens. The Royal Botanic Gardens Melbourne can be reached easily by foot, bike, car and Public transport as it is close to Melbourne CBD.

   Each Forest Therapy session allows for a maximum of 20 participants. Each Forest Therapy session lasts for two hours and is conducted by two INFTA-Certified and Accredited Forest Therapy Guides.

   Two brief online surveys - which are optional to be completed by participants - will be administered before (pre-survey) and after (post-survey) each Forest Therapy session.
   * The pre-survey contains questions about participants personal background, studies and enrolment as well as their mood and wellbeing. The pre-survey will take approximately 15-20 minutes to be completed. Participants can opt out of completing the pre-survey at any time but once they have submitted their responses, these are anonymized and deletion of this data is not feasible.
   * The post-survey contains questions about how participants perceived and enjoyed the Forest Therapy session and any changes they might notice in how they are feeling. The post-survey will take approximately 5-10 minutes to be completed. Participants can opt out of completing the post-survey at any time but once they have submitted their responses, these are anonymized and deletion of this data is not feasible.

   These surveys will help to collect important data which allows measuring how effective Forest Therapy sessions are for international students. Participants' total time commitment - Forest Therapy session plus pre- and post-survey - will be less than three hours.
3. Privacy, Confidentiality and Disclosure of Information

   Participation in this research project is confidential and will not be disclosed to others without the consent of participants. The way in which participants personally respond to questions within the surveys will be immediately de-identified.

   Data from the participants' registration and the pre- and post-surveys will initially be stored on INFTA's secure cloud-based servers (conforming to ISO 27001 international security standards). At the end of the data collection, all cloud-based data will be downloaded to a secure, off-line storage at INFTA for the statistical analyses to be performed. All cloud-based data will be deleted. All identifiable information of participants (i.e., names, phone numbers, email addresses) will be removed after having been recoded into unique numerical IDs which are stored separately from survey data. The responses of participants will remain non-identifiable. Only members of the research team (see above) will have access to the de-identified data.

   Data will be securely stored for five years after the results of the research project have been published. At the end of this storage period, the data will be deleted.

   To maintain the privacy of everyone attending the Forest Therapy session, participants are requested not share any personal information with others in their group unless explicitly allowed to do so. Particiapnts are able to share their own experiences of the Forest Therapy session with friends and family but are requested not to share other people's experience.
4. Risks

   There are no expected risks for taking part in this research project.

   Sudden, unforeseen changes in weather which may afflict participants' health, will lead to a cancellation of a Forest Therapy session. Participants' health and safety comes first!
5. Benefits

   This project will help facilitate understanding of the value of Forest Therapy as an adjunct to support the health of the international student population. Results are expected to contribute to greater understanding of the potential for implementing Forest Therapy as a Public health intervention for university students, and, in the wider sense, for Australians in general.

   The outcomes will provide valuable information about the value, applicability and effectiveness of Forest Therapy in alleviating stress and mental health issues among international students. The results will allow making recommendations how to implement Forest Therapy in future, probably in a larger and more regular way. As such, we hope that participants will consider and enjoy the physical and mental health benefits of Forest Therapy during their university studies.
6. Withdrawal

   Participants who have registered for a Forest Therapy session and wish to cancel their participation can do so. They are requested to send an email to INFTA's team using the email address smip@infta.net.

   Participants can withdraw their participation from any stage of the research project. This is possible up to the moment when they submit their survey responses. Responses will not be included in data analysis unless actively submitted by participants. Once participants have submitted their responses, their data will have been de-identified, which makes it impossible to retrieve individual responses.

   Please note that the decision to withdraw from the research project will not affect participants' relationship with their university, the researchers, or any third-party organisation.
7. Registration and Participation

Participants register their interest in the Forest Therapy sessions online at a dedicated webpage which has been set up on INFTA's cloud servers. Registration requires participants to provide their given name, family name, email address and phone number as well as the university at which they study for the purpose of being contactable. Successful registration will immediately be confirmed by email. Participants will receive a brief reminder email one to two days prior to the Forest Therapy session for which they have registered. Should a Forest Therapy session have to be cancelled or postponed, for example, due to weather-related reasons, participants will also be contacted and informed by email and/or SMS.

ELIGIBILITY:
Inclusion Criteria:

* All international students currently studying, planning to study of having completed their studies at a university in Victoria (Melbourne or regional) are eligible and invited to participate.

Exclusion Criteria:

* All domestic (Australian) students currently studying, planning to study of having completed their studies at a university in Victoria (Melbourne or regional).

Participation in this research project is voluntary.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2024-03-27 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Profile of Mood States (POMS) | 120 min (duration of standardized Forest Therapy session)
  pre/post test using psychometric instrument (POMS-16 for adults); 16 items, 5-point Likert-type scale; measuring self-reported levels of stress, anxiety and vigour

CONTACTS AND LOCATIONS:
Overall Officials: Honorary Associate Professor Dr. Dieter Kotte, Principal Investigator — International Nature and Forest Therapy Alliance
Locations (1):
- International Nature and Forest Therapy Alliance (INFTA), Newtown, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No
government policy

REFERENCES:
- See also: website of the International Nature and Forest Therapy Alliance — https://infta.net